CLINICAL TRIAL: NCT00492440
Title: A Phase I Study of Subcutaneous "CYT 107" (Interleukin-7) in Refractory Metastatic Melanoma or Renal Cell Carcinoma
Brief Title: Interleukin-7 in Treating Patients With Metastatic Melanoma or Locally Advanced or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Cytheris SA (Industry)
Collaborators: Cytheris, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-04; 07-C-0114 (Other: NCI); CLI-107-04 (Other: Cytheris)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; stage III renal cell cancer; recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — Interleukin-7; Gene Expression Profiling; Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CYT107 (r-hIL-7) (Experimental)
  Interventions: Biological: recombinant interleukin-7; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: protein expression analysis; Other: flow cytometry; Other: immunoenzyme technique; Other: immunologic technique; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: recombinant interleukin-7
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: flow cytometry
Other: immunoenzyme technique
Other: immunologic technique
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Interleukin-7 may stimulate the white blood cells to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of interleukin-7 in treating patients with metastatic melanoma or locally advanced or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of recombinant interleukin-7 (IL-7) in patients with metastatic melanoma or locally advanced or metastatic renal cell carcinoma.
* Confirm the previously documented safety profile of non-glycosylated IL-7 in these patients.
* Determine the safety of higher doses of recombinant IL-7 in these patients.
* Determine the maximum tolerated dose of recombinant IL-7 in these patients.
* Determine the biologically active dose of recombinant IL-7 in these patients.

Secondary

* Determine the pharmacokinetics and pharmacodynamics of recombinant IL-7 in these patients.
* Compare the biological and clinical effects of recombinant IL-7 with non-glycosylated IL-7 in these patients.
* Determine the potential antitumor effect of recombinant IL-7 in these patients.
* Determine the dose and administration schedule of recombinant IL-7 in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to lymphocyte count (normal lymphocyte count [CD4+ T cells > 400/mm^3] vs lymphopenic [CD4+ T cells < 400/mm^3]). Patients are assigned to 1 of 2 treatment groups.

* Group 1 (normal lymphocyte count): Patients receive recombinant interleukin-7 (IL-7) subcutaneously once a week (to determine an active dose) for up to 3 weeks in the absence of disease progression or unacceptable toxicity.
* Group 2 (lymphopenic): Patients receive recombinant IL-7 subcutaneously once a week for up to 3 weeks at one dose level below the active dose determined in group 1.

Cohorts of 3-6 patients from each group receive escalating doses of recombinant IL-7 until the maximum tolerated dose (MTD) is determined. The MTD is the defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 30 additional patients may be treated at the MTD.

Patients undergo blood and bone marrow collection periodically for pharmacokinetic, pharmacodynamic, and immunological studies. Samples are analyzed for the presence of antibodies and proteins via ELISA; CD3, CD4, and CD8 T cell counts, CD127, Ki-67, and Bcl-2 expression in CD4+ and CD8+ T cells, and CD19 B cell counts via flow cytometry; and clonal B cell proliferation via PCR and flow cytometry.

After completion of study treatment, patients are followed at 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Melanoma

    * Metastatic disease
  * Renal cell carcinoma

    * Locally advanced and unresectable disease OR metastatic disease
* Refractory to standard therapy OR ineligible to receive standard therapy
* Measurable or evaluable disease
* Previously received high-dose interleukin-2 OR have a contraindication for this treatment
* No previously untreated or unstable brain metastases
* No splenic metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* PT/PTT ≤ 1.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* AST and ALT < 2.5 times ULN
* Conjugated (Direct) bilirubin ≤ 1.25 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* LVEF ≥ 45% by cardiac stress test (e.g., stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test) for patients meeting any of the following criteria:

  * History of ECG abnormalities
  * Symptoms of cardiac ischemia
  * At least 50 years of age and over
  * Familial or personal history of heart failure
  * Previously treated with antimitotic agents susceptible to trigger heart failure
* FEV_1 > 60% of predicted (for patients with a prolonged smoking history or symptoms of respiratory dysfunction)
* No concurrent cognitive impairment or likelihood of developing cognitive impairment on study therapy
* No concurrent splenomegaly or proliferative hematologic disease
* No documented HIV positivity
* No acute hepatitis A or hepatitis B or C

  * Positive hepatitis B serology indicative of previous immunization (i.e., HBs Ab positive and HBc Ab negative) allowed
  * Positive hepatitis C serology allowed provided HCV RNA load by PCR is negative
* Resting blood pressure ≤ 140/90 mm Hg on standard antihypertensive therapy

  * Untreated hypertensive patients who received standard antihypertensive therapy allowed provided hypertension is well controlled
* No QTc prolongation ≥ 470 msec
* No prior history of cardiovascular disease, arrhythmias, or significant ECG abnormalities
* No active infection requiring systemic treatment and/or hospitalization within the past 28 days

  * Patients who have completed therapy or are clinically stable on therapy, in the opinion of the investigator, are eligible
* No history of autoimmune disease
* No history of severe asthma
* No history of medical or psychiatric disease that would preclude study treatment
* No documented cirrhosis or documented acute hepatitis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior systemic corticosteroid therapy
* More than 4 weeks since prior and no other concurrent cytotoxic therapy, immunotherapy, biological agents (i.e., cytokines, growth factors, or monoclonal antibodies), or antitumor vaccines
* More than 7 days since prior hepatotoxic drugs unless medically necessary
* More than 2 days since prior alcohol consumption
* More than 1 day since prior acetaminophen use
* No prior splenectomy
* No prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation
* No concurrent palliative therapy
* No concurrent chemotherapy
* No concurrent chronic anticoagulation (i.e., high-dose warfarin or heparin)

  * Warfarin dose 1 to 2 mg/day allowed
* No concurrent chronic medications for asthma
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety of recombinant interleukin-7 (IL-7)

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics of IL-7
Comparison of the biological and clinical effects of recombinant IL-7 with non glycosylated IL-7
Potential antitumor effect of recombinant IL-7
Dose and administration schedule of recombinant IL-7

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States